CLINICAL TRIAL: NCT01309659
Title: A Randomized, Open-Label, Wait-list Control Trial To Evaluate the Efficacy of Intravenous Iron in Older Adults With Unexplained Anemia and a Serum Ferritin Between 20 and 200 ng/mL
Brief Title: Trial To Evaluate the Efficacy of Intravenous Iron in Older Adults With Unexplained Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00028687; U01AG034661 (NIH); PACTTE_01; NCT01413919 (obsolete NCT alias)
Record Dates: First submitted 2011-02-17; First posted 2011-03-07 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Anemia; Unexplained Anemia (UAE)
Keywords: Anemia; Unexplained anemia; elderly; geriatric; older adults; UAE; over 65; iron; pactte; pactee; aging; aged; old; older
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Intervention Group (Experimental): Subjects randomized to the immediate treatment group will be scheduled to begin treatment with IV iron infusion immediately (or within 2 business days). They will receive 200mg IV iron sucrose a week for 5 weeks followed by 19 weeks of follow up.
  Interventions: Drug: iron sucrose
- Wait List Control (Experimental): Subjects randomized to the wait list control group will have an observation visit at week 6 and week 12. After that they will begin treatment with IV iron infusion. They will receive 200mg IV iron sucrose a week for 5 weeks followed by 7 weeks of follow up
  Interventions: Drug: iron sucrose

INTERVENTIONS:
Drug: iron sucrose — Patients will receive intravenous iron sucrose preparation at a dose of 200 mg per week through a peripheral intravenous catheter.
  Other Names: Venofer®
  Arms: Immediate Intervention Group
Drug: iron sucrose — Following 12 weeks of observation patients will receive intravenous iron sucrose preparation at a dose of 200 mg per week through a peripheral intravenous catheter.
  Other Names: Venofer®
  Arms: Wait List Control

SUMMARY:
The purpose of this study is to determine whether treatment of unexplained anemia in older adults with a short course of weekly intravenous iron infusions can improve physical activity and therefore quality of life.

DETAILED DESCRIPTION:
There is a tremendous morbidity and mortality associated with anemia in the elderly and the increasing proportion of elderly adults underscores the population's attributable risk of anemia. As a potentially modifiable factor, an urgent need exists to delineate the impact of anemia correction in the elderly. The Partnership for Anemia: Clinical and Translational Trials in the Elderly (PACTTE) consortium has been created to focus on treatment strategies for anemia in elderly patients. The data presented in this protocol provides a compelling rationale to evaluate the impact of a well-tolerated IV iron preparation in community dwelling older anemic adults with intermediate serum ferritin values.

Subjects will be 65 years or older adults with unexplained anemia and a serum ferritin between 20 and 200 ng/mL.

Subjects will be randomized on a 1:1 basis to either receive a 5 week course of treatment with intravenous iron immediately or to a waitlist control group who will receive treatment with intravenous iron following a 12 week observation period. Both groups will ultimately receive 200mg of intravenous iron sucrose weekly for 5 weeks to determine if this can lead to improvement in 6 Minute Walk Test results. The primary endpoint is change in 6 Minute Walk Test distances from baseline to 12 weeks. The procedures in this protocol will include the use of outcomes tools that have been selected for their ability to show improvement in quality of life in this patient population. Blood samples will also be collected for analysis both at the local lab (safety tests - eg hemoglobin or Hb) or at a central lab for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Hemoglobin concentration ≥ 9.0 g/dL and < 11.5 g/dL (women) or < 12.7 g/dL (men)
* Unexplained anemia
* Serum ferritin level ≥ 20 and ≤ 200 ng/mL
* Able to walk without the use of a walker, motorized device or the assistance of another person.
* Able to understand and willing to provide written informed consent in the absence of dementia
* Must be able to understand and speak in English

Exclusion Criteria:

* Red blood cell transfusions within the past 3 months
* Use of erythropoiesis stimulating agents (ESA) in the past 3 months
* Intravenous Iron Infusions within the past 3 months
* Distance on baseline 6MWT (6 minute walk test) above the median for age and sex
* History of unstable angina or myocardial infarction in the past 3 months
* History of stroke or TIA (transient ischemic attack) the past 3 months
* Uncontrolled hypertension (diastolic blood pressure > 100 mm Hg or systolic blood pressure > 160 mm Hg on 2 separate occasions)
* Positive fecal occult blood test within the screening period
* Elevated AST (aspartate aminotransferase) or ALT (alanine aminotransferase) ≥ 2x upper limit of normal
* Documented anaphylactic reaction to iron sucrose infusion in the past
* Subjects initiated on oral iron supplementation within the last 6 weeks, or those initiated on oral iron within the last 3 months who have had at least a one gram/dL improvement in Hb since starting oral iron supplementation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Price, MD, Principal Investigator — Stanford University MC; Stanley Schrier, MD, Study Chair — Stanford University; Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University Geriatrics Center, Baltimore, Maryland
  - Case Western Reserve University Medical Center, Cleveland, Ohio
  - Institute For Advanced Studies in Aging, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Intervention Group | Wait List Control
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Wait List Control | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
hemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.19 (0.64) | 11.3 (.80) | 11.25 (.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Test Results
Description: Subjects were asked to walk for 6 minutes, unassisted. The distance walked was recorded in meters at baseline (time of randomization) and 12 weeks after baseline (time of randomization). The change from baseline to 12 weeks, related to distance, is compared and documented.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 9
meters | 8.05 (55.48) | -11.45 (49.46)

2. Secondary Outcome: Number of Participants Who Had a Hemoglobin Increase >= 1g/dL
Description: To assess the efficacy of IV iron sucrose in improving Hemoglobin by at least 1 g/dL; an increase from baseline to week 12.
Time Frame: baseline, 12 weeks
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 10
participants | 1 | 0

3. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Trail Making Test Part B
Description: To quantify the impact of anemia treatment by IV iron sucrose on cognitive outcomes based on the Trail Making Test (TMT) Part B as measured by subjects drawing a line from 25 circled numbers to letters in 300 seconds. The change in seconds per completed circle from baseline to week 12.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. The number of participants analyzed is correct as 4 subjects for the wait list control group did not respond to this during their clinic visit.
Measure: Mean (Standard Deviation); unit: change in seconds per completed circle
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 5
change in seconds per completed circle | -0.77 (3.54) | -4.96 (8.14)

4. Secondary Outcome: Change in Self Reported Outcomes Measures as Reported by Short Form-36 (SF-36) Physical Component Score (PCS)
Description: To quantify the impact of anemia treatment by IV iron sucrose on self-reported outcomes measures by change in SF36 physical component score. The SF-36 form identifies self-report physical function and global measure of quality of life and is a multi-purpose, short-form health survey consisting of 36 questions. The Physical Component Summary (PCS) is a subscale of the SF-36 that correlates with physical health domains of the SF-36 ( Physical Function, Role-Physical, and Bodily Pain). The change is calculated and compared from baseline to week 12. The SF-36 PCS score is a norm based sore with a mean of 50 and standard deviation of 10 where results above and below 50 are above and below the average, respectively, in the 2009 general US population.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Number of participants analyzed is correct- 2 subjects for Waitlist Group did not respond.
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 8
t score | -1.89 (2.44) | -3.17 (10.95)

5. Secondary Outcome: Correlation Between Baseline Serum Ferritin, Serum Iron, and Transferrin Saturation and the Change in Hemoglobin (HB)
Description: Correlation between baseline serum ferritin, serum iron, and transferrin saturation and the change in HB from baseline to 12 weeks.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 10
correlation coefficient
  Correlation btw baseline ferritin & change in Hgb | 0.383 | 0.189
  Correlation btw baseline iron & change in Hgb | 0.323 | 0.541
  Correlation btw baseline TST & change in Hgb | 0.200 | 0.584
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.308, t-test, 2 sided — Correlation between ferritin and change in hemoglobin in the immediate intervention group. Testing the correlation equal to 0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.601, t-test, 2 sided — Correlation between ferritin and change in hemoglobin in the waitlist group. Testing the correlation = 0
Statistical Analysis 3: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.396, t-test, 2 sided — Correlation between iron and change in hemoglobin in the intermediate intervention group. Testing the correlation = 0
Statistical Analysis 4: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.106, t-test, 2 sided — Correlation between iron and change in hemoglobin in the waitlist group. Testing the correlation = 0
Statistical Analysis 5: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.606, t-test, 2 sided — Correlation between transferrin saturation and change in hemoglobin in the immediate intervention group. Testing the correlation = 0
Statistical Analysis 6: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.077, t-test, 2 sided — Correlation between transferrin saturation and change in hemoglobin in the waitlist group. Testing the correlation = 0

6. Secondary Outcome: Change in Frailty Component Related to Fatigue/ Exhaustion
Description: Subjective fatigue/exhaustion: If any of the following three criteria are met, the patient will be classified as frail for fatigue/exhaustion:
  1. "In the past month, on average, have you been feeling unusually tired during the day?" is answered "yes" and indicated as "all of the time" or "most of the time."
  2. "In the past month, on average, have you felt unusually weak?" is answered "yes" and indicated as "all of the time" or "most of the time."
  3. Energy level on a scale of 0 (no energy) to 10 (most energy) reported as ≤ 3. If the subject answers YES to any of the above noted 3 questions, then they are classified as FRAIL.
  The change in frailty for fatigue/ exhaustion is defined as changing from frail at baseline to not frail at week 12 as reported by the subject.
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Results reported by number of participants reporting change from their baseline exhaustion, and low energy.
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 10
participants
  Frailty change - self reported exhaustion | 9 | 10
  Frailty change - self-reported low energy | 0 | 0

7. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Speed of Processing
Description: To quantify the impact of anemia treatment by IV iron sucrose on cognitive outcomes based on speed of processing was derived using the z-scores of the following three tests: (1) TMT Part A seconds per completed circle, (2) simple reaction time from the CogState Detection Task, and (3) choice reaction time from the CogState Identification Task. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the subject's score at the time point from the overall baseline mean of the test and then dividing by the overall baseline standard deviation of the test. Positive z-scores indicate a better performance compared to the baseline average.
Time Frame: Baseline, 12 Week
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random.The number of participants analyzed is correct as 1 subject for the Immediate Intervention Group did not respond to this during their clinic visit.
Measure: Mean (Standard Deviation); unit: change in Z-Score
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 8 | 9
change in Z-Score | 0.62 (1.00) | 1.08 (0.88)

8. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Composite Complex Attention/Executive Processing
Description: To quantify the impact of anemia treatment by IV iron sucrose on cognitive outcomes based on Complex attention/executive processing was derived using the z-scores of the following three tests: (1) TMT Part B seconds per completed circle, (2) time score from the CogState One Back Task, and (3) accuracy score from the CogState One Back Task. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the overall baseline mean of the test from the subject's score at the time point (accuracy score) or by subtracting the subject's score at the time point from the overall baseline mean of the test (TMT and time score) and then dividing by the overall baseline standard deviation of the test.
Time Frame: Baseline, 12 week
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random.The number of participants analyzed is correct as 1 subject for the Wait List Control did not respond to this during their clinic visit.
Measure: Mean (Standard Deviation); unit: change in Z-score
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 8
change in Z-score | 0.36 (1.28) | 0.69 (1.19)

9. Secondary Outcome: Change in Cognitive Outcome Measures as Determined by Composite Learning and Memory
Description: To quantify the impact of anemia treatment by IV iron sucrose on cognitive outcomes based on Learning and memory was derived using the z-scores of the following three tests: (1) CogState ISL immediate recall score (total score from three learning trials), (2) CogState ISL immediate recall score from the first learning trial, and (3) CogState ISL delayed recall scores. The composite score for a subject at each time point was defined as the mean of the Z-scores for the three tests at the time point. For each subject, the Z-score for each test at time point was derived by subtracting the overall baseline mean of the test from the subject's score at the time point and then dividing by the overall baseline standard deviation of the test. Higher numbers indicated a better response.There is no scale, as the results are normalized variables.
Time Frame: Baseline, 12 week
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random.The number of participants analyzed is correct as 2 subjects for each of the groups did not have a response for this data.
Measure: Mean (Standard Deviation); unit: change in Z-score
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 7 | 7
change in Z-score | 0.41 (1.50) | 1.39 (2.36)

10. Secondary Outcome: Change in Self Reported Outcomes Measures as Reported by FACIT-AN Total Score
Description: To quantify the impact of anemia treatment by IV iron sucrose on self -reported outcomes measures by subjects answering 47 questions for patients with anemia and or fatigue. This test detects self-report functional changes and QoL. Change from baseline to 12 weeks. Scores range from 0-188 with higher scores indicating better function.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random.The number of participants analyzed is correct as for each of the groups there was missing responses for subjects.
Measure: Mean (Standard Deviation); unit: change in the total score
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 8 | 6
change in the total score | 10.6 (10.0) | 0.0 (34.7)

11. Secondary Outcome: Change in the Frailty Component as Determined by Self-reported Activity Level
Description: To quantify the impact of anemia treatment by IV iron sucrose on change in the frailty as measured by change in self-reported activity level. Frailty for activity level is classified by subjects responses to 6physical activity questions on the short version of the Minnesota Leisure Time Activity Questionnaire , were related to walking for exercise, moderately strenuous outdoor chores, dancing, bowling, and regular exercise. The Women's Health And Aging Study (WHAS) scoring algorithm was used to define frailty for self-reported activity level. The answers to these questions were used to calculate kilocalories (Kcals) per week, using the WHAS algorithm, which is further satisfied by by gender. For men, Kcals < 128 per week is frail. For women, Kcals < 90 per week is frail. This is a categorical measurement of yes or no. The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at week 12.
Time Frame: Baseline, 12 week
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Two subjects in the immediate intervention group and 5 subjects in the wait list group did not respond.
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 7 | 5
participants | 0 | 0

12. Secondary Outcome: Change in Frailty Component as Determined by Grip Strength
Description: To quantify the impact of anemia treatment by IV iron sucrose on change in the frailty as measured by change in grip strength. Subjects squeeze the grip strength machine 3 times with each hand. For the frailty outcome the maximum grip strength from the dominant hand is used. (change from frail at baseline to not frail at week 12). Grip strength is stratified by gender and BMI. For men with (BMI <= 24 and a grip strength (GS) <= 29) or (BMI 24.1-28 and grip strength <= 30) or (BMI >28 and a grip strength <= 32) were classified as "frail". For women with (BMI <= 23 and a grip strength of <= 17) or (BMI 23.1-26 and a GS <= 17.3) or (BMI 26.1-29 and a GS <= 18) or (BMI > 29 and a GS <= 21) were classified as "frail".The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at week 12.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Three subjects in both the immediate intervention group and the wait list control groups were missing responses.
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 6 | 7
participants | 0 | 0

13. Secondary Outcome: Change in Frailty Component as Determined by the 4 Meter Walk Speed
Description: To quantify the impact of anemia treatment by IV iron sucrose on change in the speed of the 4 meter walk speed. Subjects are asked to walk as fast as they can for 4 meters. Frailty was determined by the subject's speed. (change from frail at baseline to not frail at week 12). 4 m walking speed is stratified by gender and height. For men, (height of <= 173 cm and a walking speed of <= 0.65 meter/sec) or a (height > 173, <= .76 meter/sec) were classified as "frail". For women, (height of <= 159 cm and a walking speed of <=.65 meter/sec) or (height >159 cm <= 0.76 meter/sec) were classified as "frail".The outcome is the number of participants who were classified as "frail" at baseline and changed to "not frail" at week 12.
Time Frame: Baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Five subjects were missing responses in the immediate intervention group and four subjects were missing responses in the wait list control group.
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 4 | 6
participants | 0 | 0

14. Secondary Outcome: Correlation Between Baseline Soluble Transferrin Receptor and the Change in HB From Baseline to 12 Weeks
Description: Correlation between baseline soluble transferrin receptor and the change in hemoglobin from the baseline to 12 weeks.
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. One subject in both the immediate intervention and the wait list control groups were missing responses.
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 8 | 9
correlation coefficient | -0.192 | -0.886
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.649, t-test, 2 sided — Correlation between soluble transfer receptor and change in hemoglobin in the immediate intervention group. Testing the correlation =0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — Correlation between soluble transfer receptor and change in hemoglobin in the wait list group. Testing the correlation =0

15. Secondary Outcome: Correlation Between Baseline Soluble Transferrin Receptor Index (Soluble Receptor/Log Ferritin) and the Change in Hemoglobin
Description: Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in hemoglobin from baseline to 12 weeks.
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Four subjects were missing responses from both the immediate intervention group and the wait list control group.
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 5 | 6
correlation coefficient | -0.500 | -0.714
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.391, t-test, 2 sided — Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in hemoglobin in the immediate intervention group. Testing correlation =0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.111, t-test, 2 sided — Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in hemoglobin in the wait list control group. Testing correlation =0

16. Secondary Outcome: Correlation Between Baseline Serum Ferritin, Serum Iron, and Transferrin Saturation and the Change in 6 Minute Walk Test Distance
Description: Correlation between baseline serum ferritin, serum iron, and transferrin saturation and the change in 6 Minute Walk Test distance from baseline to 12 weeks.
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. One subject was missing responses from the wait list control group.
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 9 | 9
correlation coefficient
  Correlation for ferritin | 0.617 | 0.100
  Correlation for iron | 0.332 | -0.133
  Correlation TSAT | 0.400 | -0.350
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.077, t-test, 2 sided — Correlation between baseline serum ferritin and the change in 6 Minute Walk Test distance in the immediate intervention group. Testing correlation =0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.798, t-test, 2 sided — Correlation between baseline serum ferritin and the change in 6 Minute Walk Test distance in the wait list group. Testing correlation =0
Statistical Analysis 3: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.383, t-test, 2 sided — Correlation between baseline iron and the change in 6 Minute Walk Test distance in the immediate intervention group. Testing correlation =0
Statistical Analysis 4: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.732, t-test, 2 sided — Correlation between baseline iron and the change in 6 Minute Walk Test distance in the wait list group. Testing correlation =0
Statistical Analysis 5: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.286, t-test, 2 sided — Correlation between baseline transferrin saturation and the change in 6 Minute Walk Test distance in the immediate intervention group. Testing correlation =0
Statistical Analysis 6: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.356, t-test, 2 sided — Correlation between baseline transferrin saturation and the change in 6 Minute Walk Test distance in the wait list group. Testing correlation =0

17. Secondary Outcome: Correlation Between Baseline Soluble Transferrin Receptor and the Change in the 6 Meter Walk Test Distance
Description: Correlation between baseline soluble transferrin receptor and the change in the 6 Meter Walk Test distance from baseline to 12 weeks
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. One subject was missing responses in the immediate intervention group and one subject was missing responses in the wait list control group.
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 8 | 9
correlation coefficient | 0.192 | 0.349
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.649, t-test, 2 sided — Correlation between baseline soluble transferrin receptor and the change in the 6 Meter Walk Test distance of the immediate intervention group. Testing correlation =0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.396, t-test, 2 sided — Correlation between baseline soluble transferrin receptor and the change in the 6 Meter Walk Test distance of the wait list group. Testing correlation =0

18. Secondary Outcome: Correlation Between Baseline Soluble Transferrin Receptor Index (Soluble Receptor/Log Ferritin) and the Change in the 6 Minute Walk Test Distance
Description: Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in the 6 Minute Walk Test Distance from baseline to 12 weeks
Time Frame: baseline, 12 weeks
Population: All intent-to-treat patients were included in the primary analysis with an assumption that any missing data were missing completely at random. Four subjects were missing responses in the immediate intervention group and four subjects were missing responses in the wait list control group.
Measure: Number; unit: correlation coefficient
Arm/Group | Immediate Intervention Group | Wait List Control
Number analyzed (Participants) | 5 | 6
correlation coefficient | -0.300 | 0.486
Statistical Analysis 1: Comparison: Immediate Intervention Group; Test type: Superiority or Other; p = 0.624, t-test, 2 sided — Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in the 6 Minute Walk Test Distance in the intermediate intervention group. Testing correlation =0
Statistical Analysis 2: Comparison: Wait List Control; Test type: Superiority or Other; p = 0.329, t-test, 2 sided — Correlation between baseline soluble transferrin receptor index (soluble receptor/log ferritin) and the change in the 6 Minute Walk Test Distance in the wait list group. Testing correlation =0

ADVERSE EVENTS:
Arm/Group | Immediate Intervention Group | Wait List Control
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 7/9 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention Group (N=9) | Wait List Control (N=10)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention Group (N=9) | Wait List Control (N=10)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infecction (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 1 (1) | 0 (0)
Spinal Pain (General disorders) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No